CLINICAL TRIAL: NCT04090164
Title: Association of Hepatitis C Virus Seropositivity With Breast Cancer Prognosis and Treatment Outcome
Brief Title: Association of Hepatitis C Virus With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Osama Hussein, Professor of surgery (surgical oncology), Mansoura University
Other Study IDs: R.18.02.34.R1.R2
Record Dates: First submitted 2018-01-14; First posted 2019-09-16 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Hepatitis C
Keywords: Breast cancer; Hepatitis C virus; Prognosis; Epidemiology
MeSH Terms: conditions — Breast Neoplasms; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: The data of breast cancer patients treated at OCMU in the last 10 years will be retrieved from the hospital data filing system. All consecutive patients with biopsy-proven invasive breast cancer will be included.
- Control group: A group of age-matched women from the same geographical distribution who are healthy volunteers or hospital patients without cancer diagnosis will serve as a control group for the HCV prevalence. We aim at a sample size with a study-to-control ratio of 1:3.

SUMMARY:
Hepatitis C viral infection is a major health problem in Egypt. The management of breast cancer patients is often complicated by the presence of associated HCV infection. This study aims at investigating the epidemiological association of the two conditions. It will also investigate the possible correlation with treatment outcome.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in adult Egyptian females. The world's highest prevalence of hepatitis C virus is found in Egypt. Several investigators examined the epidemiological association of HCV with breast cancer. Published literature reports conflicting results regarding the HCV association with breast cancer incidence. Population-based studies from HCV-endemic area demonstrated increased breast cancer incidence in HCV-positive women younger than 50 years. On the other hand, population studies from HCV-low prevalence regions failed to detect an association of the virus with breast cancer.

HCV seropositive patients constitute a large sector of oncology patients treated in Egyptian practice. HCV infection with or without clinically-significant liver disease impose several therapeutic, social and logistic problems. Recently, investigators from Mansoura University reported their findings among breast cancerpatients. According to these data, HCV-positive breast cancer patients had several markers of disease aggression such as large tumor size, high tumor grade and nodal infiltration. Moreover, HCV-NS4 (non-structural protein-4) blood levels positively correlated with the level of the known breast cancer marker CA15-3.

In the current study, the investigators will investigate the incidence of HCV seropositivity in breast cancer patients and an age-matched control group. The study also examines the association of HCV status on the patients' baseline characteristics such as tumor stage and grade and with patients' treatment plan and treatment outcome.

Specifically, the aims of the study are the following:

1. To test if HCV seropositivity is associated with breast cancer diagnosis in Egyptian population.
2. To test if HCV-positive patients harbour more aggressive breast tumors.
3. To test if HCV-positivity affects management decision in breast cancer patients.
4. To test if HCV-positive patients suffer more frequent adverse effects to breast cancer treatment.
5. To compare disease-free survival of HCV seropositive breast cancer patients vs. seronegative patients.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven invasive breast cancer.

Exclusion Criteria:

* Patients with unknown viral marker status.
* Patients who did not complete their management at OCMU.
* Patients with multiple cancer diagnoses.
* Patients with virus-unrelated hepatic pathology.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of all consecuitive patients on Oncology Center of Mansoura University (OCMU) database.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Oncology Center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Su FH, Chang SN, Chen PC, Sung FC, Su CT, Yeh CC. Association between chronic viral hepatitis infection and breast cancer risk: a nationwide population-based case-control study. BMC Cancer. 2011 Nov 24;11:495. doi: 10.1186/1471-2407-11-495. PMID 22115285
- [Background] Attallah AM, El-Far M, Abdelrazek MA, Omran MM, Mahmoud AZ, Khalifa HS, Ahmed MM, El-Dosoky I. HCV nonstructural protein 4 is associated with aggressiveness features of breast cancer. Breast Cancer. 2018 May;25(3):297-302. doi: 10.1007/s12282-017-0829-1. Epub 2017 Dec 28. PMID 29285674
- [Background] El-Ghitany EM, Farghaly AG. Geospatial epidemiology of hepatitis C infection in Egypt 2017 by governorate. Heliyon. 2019 Aug 17;5(8):e02249. doi: 10.1016/j.heliyon.2019.e02249. eCollection 2019 Aug. PMID 31463388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Hospital medical record system was searched to identify patients with the "malignant neoplasm of the breast" diagnosis. The information of an un-selected sample of 650 patients was retrieved from the system. Two-hundred forty-five patients with incomplete data were excluded. The remaining 405 patients were subjected for further analysis.
Pre-assignment Details: The study group was retrospectively extracted from hospital file. However, The "Dakahlia Governorate adult female Population" is a historical control group derived from the raw data of a previous study. As such, this control group has not been recruited in the current study.
Groups:
- Dakahlia Governorate Adult Female Population: One-hundred forty-five adult females from Dakahlia governorate were sampled in a published population-based cross sectional study from 2015 to 2017.
  [El-Ghitany EM, Farghaly AG (2019) Geospatial epidemiology of hepatitis C infection in Egypt 2017 by governorate. Heliyon 5 (8):e02249. doi:10.1016/j.heliyon.2019.e02249}
Period: Overall Study
Arm/Group | Study Group | Dakahlia Governorate Adult Female Population
Started | 650 (Number of patients retrivied from the hospital files.) | 145
Completed | 405 (Number of patients analyzed.) | 145
Not Completed | 245 | 0
Not completed — incomplete data on file | 245 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Group: Randomly selected data of 405 patients treated within the last ten years at the study site.
- Dakahlia Governorate Adult Female Population: A historical control group derived from the raw data of a previously published study (PMID: 31463388, PMCID: PMC6709406, DOI: 10.1016/j.heliyon.2019.e02249)
- Total: Total of all reporting groups
Arm/Group | Study Group | Dakahlia Governorate Adult Female Population | Total
Number analyzed (Participants) | 405 | 145 | 550
Age, Customized [Count of Participants; unit: Participants]
  < 45 years | 127 | 93 | 220
  45 years or above | 278 | 52 | 330
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 405 | 145 | 550
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 405 | 145 | 550

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of HCV Seropositivity in Breast Cancer Patients.
Description: Percentage of patients with breast cancer with positive anti-HCV serological test.
Time Frame: This outcome will be assessed through study completion, an average of 6 months.
Measure: Count of Participants; unit: Participants
Groups:
- Dakahlia Governorate Adult Female Population: One-hundred forty-five adult females from Dakahlia governorate were sampled in a published population-based cross sectional study from 2015 to 2017.
Arm/Group | Study Group | Dakahlia Governorate Adult Female Population
Number analyzed (Participants) | 405 | 145
Participants
  anti-HCV Seropositive | 88 | 15
  anti-HCV seronegative | 317 | 130
Statistical Analysis 1: Comparison: Study Group vs Dakahlia Governorate Adult Female Population; Fisher exact test was used for testing of association of Breast Cancer diagnosis with anti-HCV test status; Test type: Other; p = 0.0027, Fisher Exact; Odds Ratio (OR) = 2.406, 95% CI 2-sided [1.341 to 4.316]
Statistical Analysis 2: Comparison: Study Group vs Dakahlia Governorate Adult Female Population; Fisher exact test was used to test the association of Breast Cancer diagnosis with anti-HCV test result in women younger than 45 years; Test type: Other; p = 0.0034, Fisher Exact; Odds Ratio (OR) = 7.032, 95% CI 2-sided [1.582 to 31.25]

2. Secondary Outcome: Disease-related Events
Description: The number of events related to breast cancer diagnosis. Disease-free survival (DFS) was calculated as the time from the date of breast cancer diagnosis to the date of last follow-up or the date of first breast cancer-related event. At the time of analysis, median survival has not been reached.
Time Frame: at the date of last patients' visit recorded on her file. Patients should be censored at least 12 months from the time of diagnosis.
Population: At the time of analysis, median survival has not been reached. This Outcome Measure was pre-specified to be collected only for the Study Group. The outcome is not applicable to the control group (non-cancer population).
Measure: Number; unit: number of events related to cancer
Groups:
- Anti-HCV Positive Patients: patients with anti-HCV positive test.
- Anti-HCV Negative Patients: patients with anti-HCV negative test.
Arm/Group | Anti-HCV Positive Patients | Anti-HCV Negative Patients
Number analyzed (Participants) | 88 | 317
number of events related to cancer | 37 | 6

ADVERSE EVENTS:
Time Frame: All-cause Mortality and Adverse Events were not assessed in this Retrospective, observational study.
Description: All-cause Mortality and Adverse Events were not assessed in this retrospective, observational study
Groups:
- Study Group: All-cause Mortality and Adverse Events were not assessed in this retrospective, observational study
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This is a retrospective study. Due to limited funding, a non-selected sample of Breast Cancer was compared to a historical control derived from the data of a previously published population study. Further studies are required.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT04090164/Prot_SAP_000.pdf